CLINICAL TRIAL: NCT02623647
Title: A Phase I-II Study on the Tolerance and Efficacy of SBRT in 3 Fractions for Low/Int Risk Prostate Cancer
Brief Title: A Phase I-II Study on Stereotactic Body Radiotherapy in 3 Fractions for Low/Int Risk Prostate Cancer
Acronym: eHYPO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: San Giovanni Addolorata Hospital (Other); Azienda Sanitaria-Universitaria Integrata di Udine (Other)
Responsible Party: Principal Investigator, Giuseppe Sanguineti, Chairman, Dept of Radiation Oncology, Regina Elena Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eHYPO
Record Dates: First submitted 2015-12-03; First posted 2015-12-08 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A single-arm, nonrandomized (Other): stereotactic body radiotherapy SBRT, 40 Gy for 3 fractions
  Interventions: Radiation: stereotactic body radiotherapy SBRT

INTERVENTIONS:
Radiation: stereotactic body radiotherapy SBRT — 40 Gy in 3 fractions to the prostate gland delivered with stereotactic body radiotherapy

SUMMARY:
The present is a phase I-II study testing the safety and the efficacy of extremely hypofractionated radiotherapy for early stage prostate cancer. The study is designed to assess GU toxicity while controlling tumor control, in terms of survival free from biochemical failure. 40 Gy in fxs will be delivered to patients with low and favourable intermediate risk prostate tumors.

DETAILED DESCRIPTION:
In the last two decades several studies have shown an exclusive sensitivity of prostate cancer cells to low doses per fraction. It has been postulated that the effect of fractionation is protective against tumor cells rather than both acute and late responding normal tissues, and this in turn tends to decrease the therapeutic index. The schedule tested here is considered biologically equivalent to deliver to the tumor, at 2 Gy per fraction, a total dose of approximately 170 Gy or more than twice of the reference schedule (76-80 Gy). On the contrary, the schedule is considered to deliver a dose of 78 Gy and 130 Gy on acute (i.e mucosa)(a/b =10 Gy) and late (a/b =3 Gy)(i.e. rectum, bladder) responding tissues.

Main selection criteria: Patients (>18 yrs/old) with low risk (primary tumor stage according to AJCC 2010: T1-2a and Gleason Score-GLS: 3+3 and serum Prostate Specific Antigen-PSA: PSA<10 ng/ml) and among those with intermediate risk features (clinical stage T2b-c or GLS 7 or PSA of 10-20 ng/ml) those with favorable ones (a single factor for intermediate risk and GLS 3 + 4 and <50% of biopsy cores containing cancer) will be selected.

Work up & pretreatment procedures: A diagnostic biopsy with at least 10 cores is needed. Patients will undergo in local anesthesia the placement both 4 fiducials (or 'gold seeds') and a gel spacer between the prostate and the rectum at least one week before the simulation. Both the seeks and the gel spacer are implanted throughout the perineum. The gel will be inserted between the posterior aspect the prostate and the anterior rectal wall to obtain a space of at least 5 mm in thickness between the two structures.

Treatment outline: Patients will be treated with EBRT, Volumetric Arc Radiotherapy on the prostate only to the total dose of 40 Gy in 3 fractions, every other day (dose per fraction=13.3 Gy). While neoadjuvant androgen deprivation is allowed for up to 3 months, no concomitant/adjuvant (to eHYPO) androgen deprivation is allowed.

Simulation & Planning: Patients will undergo both CT and MR of the pelvis for planning purposes, in the supine position.

The clinical target volume (CTV) is represented by the prostate as identified on MR images (coregistered with the CT). During both CT and MR scans the patient will be catheterized (to identify the urethra) and the bladder filled with saline, 250 cc. The prostate (target) will be contoured on the MR and expanded by 4 mm isotropically for planning purposes to obtain the Planning Target Volume (PTV). The rectal wall, bladder wall, bladder trigone, prostate urethra, intestinal cavity, rectal spacer, penile bulb, femoral heads will be contoured as well. The treatment will be planned with Volumetric Arc Modulated Therapy. Before each treatment fraction, the correct set up of the prostate will be done comparing the spatial position of the 4 fiducials on the planning CT and the CBCT. Patients will be seen at each treatment, one month after treatment completion and every three months afterwards for up to 2 yrs. Serum PSA will be obtained at each follow up after treatment. Regarding disease control, outcome will computed in terms of biochemical control free survival, or survival with biochemical control. This will defined according to the 'Phoenix' definition of 'nadir plus 2 ng/ml'. Toxicity will be recorded with CTCAE v4.0 at each examination. Before treatment and at both 12 and 24 month follow ups patients will report QoL (EORTC and FACT-P), IPSS, urinary continence (ICIQ-SF) and sexual activity (IIEFS). At 12 and 24 months they will be asked to report satisfaction with treatment (FACIT-I).

ELIGIBILITY:
Inclusion Criteria:

* age (>18 yrs/old)
* low risk prostate cancer defined as primary tumor stage according to AJCC 2010: T1-2a and Gleason Score-GLS: 3+3 and serum Prostate Specific Antigen-PSA: PSA<10 ng/ml); or among intermediate risk prostate cancer defined as clinical stage T2b-c or GLS 7 or PSA of 10-20 ng/ml, only patients with favourable characteristics: a single factor for intermediate risk AND GLS 3 + 4 AND <50% of biopsy cores containing cancer (12 cores as a minimum).

Exclusion Criteria:

* prior radiotherapy
* concomitant androgen deprivation
* pt failure to consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-03 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
grade 2+ GU toxicity according to CTCv4.0 | 1 yr
  Hematuria (A disorder characterized by laboratory test results that indicate blood in the urine) Urinary incontinence ( A disorder characterized by inability to control the flow of urine from the bladder.)

SECONDARY OUTCOMES:
biochemical failure according to Phoenix definition (nadir + 2 ng/ml) | 5-yr
  A prostate specific antigen (PSA) cutoff point of 0.2 ng./ml. has been suggested as the standard definition of disease freedom for curative treatment of localized prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Sanguineti, MD, Principal Investigator — Regina Elena National Cancer Institute, Rome IT
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: No